CLINICAL TRIAL: NCT06907251
Title: Dapagliflozin for Long COVID Syndrome
Acronym: DALCO
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Ottawa Heart Institute Research Corporation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2024OCT9
Record Dates: First submitted 2025-03-31; First posted 2025-04-02 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: COVID - 19; Long COVID Syndrome
Keywords: Covid-19; Long Covid syndrome; sars cov-2
MeSH Terms: conditions — COVID-19 | interventions — dapagliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Interventional (Experimental): Participants will receive 10mg dapagliflozin orally for 12 months
  Interventions: Drug: Dapagliflozin (DAPA)
- Placebo (Placebo Comparator): Participants will receive a placebo once daily for 12 months.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dapagliflozin (DAPA) — Dapagliflozin 10mg orally once a day for 12 months
  Arms: Interventional
Drug: Placebo — Participants will receive a matching placebo taken once daily by mouth for 12 months.
  Arms: Placebo

SUMMARY:
This is a randomized, placebo-controlled study. Patients with long COVID will be randomized to receive dapagliflozin or placebo for 12 months.

DETAILED DESCRIPTION:
This is a multi-centre, randomized, placebo-controlled trial (Figure 4). We will randomly assign patients with long COVID to 12 months of dapagliflozin 10 mg or placebo daily. The 10 mg daily dose of dapagliflozin was used in large clinical trials (44,48) and is the Health Canada approved dose for heart and kidney disease. Additionally, this dose was used in the MRI study of body composition (58) and the RCT in patients with acute COVID-19 (54).

Eligible patients with long COVID will be recruited from post COVID programs or advertisement through-multi-media. A total of 192 participants will be enrolled and this is anticipated to take 3 years. Participants will be followed for the entire duration of the study. Based on a study duration of 5 years (3-year recruitment, 2-year follow-up), patients will be followed for a median of 3.5 years.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older and willing and able to provide informed consent
* Patients with a history of positive COVID-19 test (polymerase chain reaction or rapid test) or have been diagnosed with COVID-19 by a health care provider.
* New or persistent symptoms at least 12 weeks from infection and present for at least 8 weeks that is not explained by an alternative diagnosis (64).
* Women of childbearing potential (WOCBP) who, if sexually active, are willing to use to use at least one highly effective methods of contraception throughout the study.

Exclusion Criteria:

* History of diabetes
* Prior heart failure
* Weight loss treatment with glucagon-like peptide-1 receptor agonists (e.g. liraglutide, semaglutide)
* Pregnancy or planned pregnancy in the next 12 months. We will ask WOCBP about the possibility of pregnancy at the time of screening and if so, then pregnancy testing will be offered. If testing is declined in this instance, then they will be excluded from the study.
* Women who are breastfeeding
* Severe renal impairment (eGFR<30mL/min1.73m2)
* Known history of allergy or hypersensitivity to dapagliflozin

Exclusion for optional MRI portion of the protocol:

- Any contraindication to MRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2028-06-30 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
6 month change in EQ-5D derived utility score. | 6 months
  The 6 month change in EQ-5D derived utility score will be compared between the dapagliflozin and placebo arms within a multiple regression model.

SECONDARY OUTCOMES:
Incident diabetes | 12 months
  New diagnosis of diabetes mellitus (fasting glucose >7.0 mmol/L. HbA!c >6.5%, new prescription of diabetes pharmacotherapy)
Cardiovascular Event | 12 months
  Cardiovascular event - atrial fibrillation, ventricular tachycardia/fibrillation, acute coronary syndrome, heart failure, transient ischemic attack, stroke, cardiovascular death

CONTACTS AND LOCATIONS:
Locations (1):
- University of Ottawa Heart Institute, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided